CLINICAL TRIAL: NCT05047562
Title: Effect of Pilates Method and Segmental Stabilization in Elderly People With Chronic Non-specific Low Back Pain: Randomized Clinical Trial
Brief Title: Effect of Pilates and Segmental Stabilization in Elderly People With Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3270664
Record Dates: First submitted 2021-09-08; First posted 2021-09-17 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-08

CONDITIONS: Low Back Pain
Keywords: Chronic Pain; Exercise Therapy; Physical Therapy Modalities
MeSH Terms: conditions — Low Back Pain; Chronic Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates Group (Active Comparator): Participants will undergo 16 sessions, twice a week on alternate days through the following Pilates Method exercises: Pelvic Curl, Leg lift Supine, One leg circle modified and Hundred modified. There will be 4 sets of 5 repetitions in the first week, 6 repetitions in the second week, 7 repetitions in the third week, 8 repetitions in the fourth week, 9 repetitions in the fifth week, 10 repetitions in the sixth to eighth week.
  Interventions: Other: Pilates Group
- Segmental Stabilization Group (Active Comparator): Participants will undergo 16 consultations, twice a week on alternate days through the following Segmental Stabilization exercises: multifidus in prone position, transverse abdomen in four supports, transverse abdomen in dorsal decubitus and transverse abdomen associated with multifidus in position orthostatic. There will be 4 sets of 10 repetitions of 10 seconds in all appointments.
  Interventions: Other: Segmental Stabilization group

INTERVENTIONS:
Other: Pilates Group — 16 Pilates exercise sessions twice a week for 2 months.
  Arms: Pilates Group
Other: Segmental Stabilization group — 16 sessions of segmental stabilization exercises, 2 times a week for 2 months.
  Arms: Segmental Stabilization Group

SUMMARY:
INTRODUCTION: Low back pain is an important health condition with great consequences from the socioeconomic point of view and is associated with high costs for the health system, absenteeism at work and reduced functional performance. It is considered one of the most relevant health problems in the elderly, with point prevalence estimates higher than for other musculoskeletal conditions. It can be defined as any pain between the last ribs and the lower gluteal folds, with or without pain in the lower limbs, manifesting itself acutely, subacutely or chronically. OBJECTIVE: To compare the effect of the Pilates method versus segmental stabilization in elderly people with chronic low back pain. METHOD: 60 elderly people with chronic low back pain will participate in the study and will be randomized into two groups: Pilates Group (GP) and Segmental Stabilization Group (SG). The two treatments will have 16 individual sessions, twice a week. Pain will be assessed using the visual analogue pain scale; functional disability, using the Oswestry disability index; excessive fear of movement and physical activity, by the Tampa scale of kinesiophobia; level of confidence in the balance for specific activities, by the ABC scale and; activation of the transversus abdominis muscle by pressure biofeedback. Individuals will be evaluated in four moments: before the first session, after the last session, three and six months after the end of the treatment to verify the effects in the medium term. Patient allocation and assessments will be performed by a blind examiner. Data will be analyzed using the ANOVA procedure and Tukey's Multiple Comparison test. The significance level will be 5%. A hipótese deste estudo é que o grupo que realiza exercícios de Pilates obtém ganhos mais obtem que o grupo que realiza exercícios de estabilização segmentar em todas as variáveis ao final do tratamento.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific low back pain for at least 3 months.
* Intensity of pain equal to or greater than 3 cm.

Exclusion Criteria:

* Specific low back pain.
* Neurological involvement (radiculopathy, myelopathy).
* Previous spinal surgery.
* Any impediment to performing the exercises.
* Having had recent surgeries.
* Being on treatment for low back pain
* Not having cognitive ability to perform the exercises or be submitted to the proposed assessments
* Missing appointments three times in a row.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-06-13 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in pain on the Numerical Pain Scale at week 16, 3 and 6 months after the end of treatment | Baseline, week 16, 3 and 6 months after completion of treatment.
  The Numerical Pain Scale is a scale from 0 to 10, with 0 meaning total absence of pain and 10 the maximum bearable pain level by the patient.
  Change = Baseline, week 16, 3 and 6 months after the end of treatment.
Change from baseline in functional disability on the Oswestry Disability Index at week 16, 3, and 6 months after the end of treatment | Baseline, week 16, 3 and 6 months after completion of treatment.
  The Oswestry Disability Index is a validated instrument for the Portuguese language with high reliability for a Brazilian population. The index is calculated by adding the total score (each section is from 0 to 5) and the total points equal to the sum of the points of the 10 sections. Interpretation is performed by means of percentage: 0% to 20% minimal disability, 21% to 40% moderate disability, 41% to 60% severe disability, 61% to 80% disability, 81% to 100% patient bedridden or exaggerating symptoms.

SECONDARY OUTCOMES:
Change from baseline to Kinesiophobia on the Tampa Kinesiophobia Scale at week 16, 3, and 6 months after the end of treatment. | Baseline, week 16, 3 and 6 months after completion of treatment.
  The Tampa scale of kinesiophobia consists of a self-administered questionnaire consisting of 17 questions that address pain and symptom intensity. The scores range from 1 to 4, with the answer "strongly disagree" equaling 1 point, "partially disagree" with 2 points, "partially agree" with 3 points, "strongly agree" with 4 points. To obtain the final total score, it is necessary to invert the scores of questions 4, 8, 12 and 16. The final score can be a minimum of 17 and a maximum of 68 points, the higher the score, the higher the degree of kinesiophobia
Change from baseline for confidence in balance to specific activities on the Activities-Specific Balance Confidence Scale at week 16, 3, and 6 months after the end of treatment. | Baseline, week 16, 3 and 6 months after completion of treatment.
  The ABC scale - Activities-Specific Balance Confidence or Confidence in Balance for Specific Activities was developed to numerically quantify the level of confidence in carrying out specific activities without losing balance or becoming unstable. The higher the score, the greater the confidence to perform the activities.
Change from baseline to transversus abdominis muscle activation in the pressure biofeedback unit at 16 weeks, 3 and 6 months after the end of treatment. | Baseline, week 16, 3 and 6 months after completion of treatment.
  The pressure biofeedback unit is a reliable instrument for the analysis of transversus abdominis muscle contraction. The lower the pressure, the greater the ability to activate this muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Ariela Cruz, Principal Investigator — University of Sao Paulo; Amelia Marques, Study Director — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, Brazil